CLINICAL TRIAL: NCT06687928
Title: A Randomized, Double-blind, Two-arm, Parallel-group, Single-dose, Phase 1 Study to Compare the Pharmacokinetics, Safety, and Immunogenicity of Subcutaneous CT-P6 and Herceptin in Healthy Male Subjects
Brief Title: To Compare the Pharmacokinetics, Safety, and Immunogenicity of Subcutaneous CT-P6 and Herceptin in Healthy Male Subjects (Trastuzumab)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-P6 1.6
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-blind, Two-arm, Parallel-group, Single-dose, Phase 1 Study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcutaneous CT-P6 (Experimental): Subcutaneous CT-P6 (CT-P6 SC): 600 mg/5 mL
  Interventions: Biological: CT-P6 SC
- Subcutaneous EU-approved Herceptin (Active Comparator): Subcutaneous Herceptin (EU-approved Herceptin SC): 600 mg/5 mL
  Interventions: Biological: EU-Approved Herceptin SC

INTERVENTIONS:
Biological: CT-P6 SC — A single fixed dose (600 mg) of CT-P6 subcutaneous
  Arms: Subcutaneous CT-P6
Biological: EU-Approved Herceptin SC — A single fixed dose (600 mg) of EU-approved Herceptin subcutaneous
  Arms: Subcutaneous EU-approved Herceptin

SUMMARY:
A Randomized, Double-blind, Two-arm, Parallel-group, Single-dose, Phase 1 Study to Compare the Pharmacokinetics, Safety, and Immunogenicity of Subcutaneous CT-P6 and Herceptin in Healthy Male Subjects

DETAILED DESCRIPTION:
CT-P6 SC, containing the active substance trastuzumab in combination with rHuPH20, is being developed by CELLTRION, Inc. (hereafter, the Sponsor) as a proposed biosimilar to the reference product, EU-approved Herceptin SC. The primary amino acid sequences of trastuzumab in CT-P6 SC are identical to those of the reference drug (EU-approved Herceptin SC). The CT P6 drug product will have the same pharmaceutical liquid formulation form and strength as the reference product's vial for SC injection and is intended to have a highly similar quality profile to the reference product.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject between 19 and 55 years of age
2. Body weight between 60 and 90 kg, BMI between 18.0 and 29.9 kg/m2
3. Subject is informed and able to understand the full nature and purpose of the study, including possible risks and side effects, and is given ample time and opportunity to read and understand this information. The subject has the ability and agrees to cooperate with the investigator and must sign and date the written informed consent prior to performing any of the Screening procedures.
4. Subject who is sexually active with a woman of childbearing potential must agree to use a highly effective and medically acceptable methods of contraception consistent with local regulations during the course of the study and for 7 months after administration of the study drug (Day 1). Examples include the following:

   1. Condom with or without spermicide
   2. True abstinence, when this is in line with the preferred and usual lifestyle of the subject
   3. Or, a female partner with hormonal contraceptive or barrier method

Subject who has been surgically sterilized for less than 24 weeks prior to the date of informed consent and his female partner of childbearing potential must agree to use any medically acceptable methods of contraception.

Exclusion Criteria:

* A medical history and/or condition that is considered significant
* Clinically significant allergic reactions, hypersensitivity
* History or congestive heart failure, NYHA class ≥ class II
* Current infection of hepatitis B virus, hepatitis C virus, human immunodeficiency virus, or syphilis
* History or current of malignancy
* Previous exposure to trastuzumab or any drugs including Human epidermal growth factor receptor 2 (HER2) targeted monoclonal antibodies
* History or current use of recombinant human hyaluronidase (rHuPH20) or drugs including rHuPH20

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-08-05 (Estimated)

PRIMARY OUTCOMES:
Demonstrate PK similarity | Up to Day 64
  maximum serum concentration (Cmax) of CT-P6 SC to EU-approved Herceptin SC
Demonstrate PK similarity | Up to Day 64
  area under the concentration-time curve from time zero to infinity (AUC0-inf) of CT-P6 SC to EU-approved Herceptin SC

CONTACTS AND LOCATIONS:
Overall Officials: Minji Ma, Study Chair — Celltrion, Inc.
Locations (1):
- Celltrion, Yeonsu-gu, Incheon, South Korea